CLINICAL TRIAL: NCT06704230
Title: Multimedia Patient Entertainment During Vascular Surgery Procedures in Regional Anesthesia
Brief Title: Stress Reduction Using Video Googles on Patients Undergoing Vascular Surgery
Acronym: MEP-VASC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Augsburg (Other)
Collaborators: HappyMed GmbH (Wien, Austria) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-1199
Record Dates: First submitted 2024-09-25; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Carotid Artery Diseases; Regional Anesthesia; Distress, Procedural
Keywords: video googles; carotid endarterectomy; distress in patients; vascular surgery
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (+ video googles) (Experimental): Patients undergoging surgery, video googles are used during surgery to reduce patient distress
  Interventions: Device: video googles
- Control group (- video googles) (No Intervention): Patients undergo surgery in the same way, no video googles or other devices for the reduction of distress is used

INTERVENTIONS:
Device: video googles — Patients undergoing surgery use video googles and a headphone to distract from surgery
  Other Names: multimedial distraction
  Arms: Intervention group (+ video googles)

SUMMARY:
One treatment option of internal carotid artery stenosis is open surgical endarterectomy. The operation is frequently carried out under regional plexus anesthesia, allowing the patient to remain awake during the procedure. This approach offers the advantage of monitoring for neurological changes during carotid artery clamping, allowing the surgical team to immediately respond by placing a shunt to ensure cerebral perfusion. As a result, performing surgery under regional anesthesia provides therefor a benefit. However, for patients, the procedure, which can last up to two hours or longer in some cases, may pose a significant burden. The fixed position, inability to move, sterile drapes over the face, manipulation by the surgical team, and anxiety about potential complications are just a few of the factors that may distress patients during the operation. Increased sweating and reports of substantial subjective distress are not uncommon if the procedure is performed under local anesthesia.

In many medical fields, devices and therapies are now being utilized to reduce patient stress in the perioperative setting. In procedures performed under local or regional anesthesia, such as in orthopedics or dentistry, efforts are being made to make operations more tolerable and less stressful for patients. For example, music and video goggles are employed to entertain and distract patients during the intervention. Newer approaches using video googles appear in more and more fields to reduce distress. Especially in vascular surgery and particularly in carotid surgery, the use of audiovisual distraction during the procedure has not been implemented to our knowledge, and its benefits remain undocumented. Because of the special setting and burden for the patients it is highly necessary to test these devices in carotid surgery and explore potential benefits for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Planed carotid endarterectomy in local anesthesia

Exclusion Criteria:

* patients which are not able to communicate because of stroke or language barrier,
* Dementia or neurological damage which impairs answering questionnaires or the understanding of the situation during surgery
* medication with steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-09 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Bloodserum cortisol levels | Cortisol levels are measured six times the day the procedure is performed. Starting at 6:30am, Arraiving at the OR, dermal incision, clamping the carotid artery, dermal suture, one hour after leaving the OR
  cortisol levels in the blood are measured on six specific times in the perioperative setting
Heartrate | The heartrate is measured six times the day the procedure is performed. Starting at 6:30am, arraiving at the OR, dermal incision, clamping the carotid artery, dermal suture, one hour after leaving the OR
  The heart rate is measured on six specific times in the perioperative setting
short questionnaire on current stress | The questionnaire is asked six times the day the procedure is performed. Starting at 6:30am, arraiving at the OR, dermal incision, clamping the carotid artery, dermal suture, one hour after leaving the OR
  The short questionnaire on current stress; is measured on six specific times in the perioperative setting.
  It is a validated score to measure actual stress, there are 6 items, with 6 a scale one to six.
  The minimal score is 6 (low distress) and 36 (high distress)
Richmond Agitation-Sedation Scale (RASS) | RASS is measured six times the day the procedure is performed.Starting at 6:30am, arraiving at the OR, dermal incision, clamping the carotid artery, dermal suture, one hour after leaving the OR
  TheRichmond Agitation-Sedation Scale (RASS) is measured on six specific times in the perioperative setting.
  It is a score typically used in anesthesia to measure agitation and sedation. The scale is from +4 (aggressive) over 0 (awake and calm) to -5 (deeply sleeping, not awakable)
Spielberger State-Trait Anxiety Inventory (STAI) | One Day. Day before surgery
  This questionnaire ist is used to measure general and anxiety related to the current situation (upcoming surgery) Used are two questionnaires with 20 items each, after recoding the answers there is a numeric value for each questionnaire. High values suggest a high feeling of fear, low values, a low feeling of fear.
Satisfaction (patient, surgeon, anesthesia) | One day. After surgery, within the next 24 hours
  After completing the surgery, all participation parties (patient, surgery and anesthesia) are asked to rate the surgery regarding to calmness of the patient, pain and distress. A numeric rating scale (0-10) is used.
Next time again? | One day. After surgery, within the next 24 hours
  Patients in the interventional group are asked, if the would like to use the video googles again in case of an other surgery
pain, distress, nervousness, fear | Questions are asked six times the day the procedure is performed.Starting at 6:30am, arraiving at the OR, dermal incision, clamping the carotid artery, dermal suture, one hour after leaving the OR
  patients are asked if the feel one of the above (using no [1] - rather no [2] - not sure [3] - rather yes [4] - yes[5]) six specific times in the perioperative setting. For each quality (pain, distress, nervousness, fear) there is measured an individual value

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Hyhlik-Dürr, Prof. Dr., Study Director — Vascular Surgery Faculty of Medicine University of Augsburg, Stenglinstr. 2 86156 Augsburg
Locations (1):
- Universitätsklinikum Augsburg, Augsburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kerndl H, Millian TP, Gurtler K, Hyhlik-Duerr A. Measuring Stress Reduction in Patients Receiving Multimedia Entertainment During Vascular Surgery Under Regional Anesthesia: Protocol for a Randomized Controlled Study. JMIR Res Protoc. 2025 Jul 11;14:e70597. doi: 10.2196/70597. PMID 40644688